CLINICAL TRIAL: NCT00672100
Title: The Effect Of Initial Local Anesthetic Dose With Continuous Interscalene Analgesia On Postoperative Pain And Diaphragmatic Function In Arthroscopic Shoulder Surgery Patients: A Double-Blind, Randomized, Parallel Group, Dose-Ranging Study
Brief Title: Initial Local Anesthetic Dose With Continuous Interscalene Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: Beaumont Foundation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIC 2007-198
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2013-05-23 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2013-05

CONDITIONS: Post-operative Pain
Keywords: Peripheral Nerve Infusion,; continuous brachial plexus block,; post-operative pain; diaphragmatic paresis
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Initial Bolus 5 ml Ropivacaine
  Interventions: Drug: Ropivacaine
- B (Active Comparator): Initial Bolus 10 ml Ropivacaine
  Interventions: Drug: Ropivacaine
- C (Active Comparator): Initial Bolus 20 ml Ropivacaine
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Initial Bolus 5 ml Ropivacaine via interscalene injection
  Arms: A
Drug: Ropivacaine — Initial Bolus 10 ml Ropivacaine via interscalene injection
  Arms: B
Drug: Ropivacaine — Initial Bolus 20 ml Ropivacaine via interscalene injection
  Arms: C

SUMMARY:
Objective: To determine a minimally effective initial local anesthetic bolus required to provide satisfactory analgesia using continuous brachial plexus infusion following arthroscopic shoulder surgery using a double-blind, randomized, study comparing 3 initial doses.

DETAILED DESCRIPTION:
Aims:

1. To compare pain ratings and supplemental analgesic requirements at discharge from PACU, 24 hours, and 48 hours and 12 weeks following 5, 10, and 20 ml boluses.
2. To compare adverse events including clinical dysphonia, Horner's syndrome, dyspnea, unexpected hospitalization, evidence of local anesthetic toxicity, and hand weakness at discharge from PACU following 5, 10, and 20 ml boluses.
3. To compare impairment in diaphragmatic excursion at discharge from PACU following 5, 10, and 20 ml boluses.
4. To compare patients' satisfaction with analgesia at 24 and 48 hours following 5, 10, and 20 ml boluses.
5. To compare patient rating of functional outcome at baseline and at 12 weeks following 5, 10, and 20 ml boluses.
6. To compare the rate of general anesthesia required following 5, 10, and 20 ml boluses.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to participation in the study.
* Is scheduled to undergo Arthroscopic Rotator Cuff Repair, defined as arthroscopically assisted repair of any of the muscles or tendons comprising the rotator cuff.
* If subject is a female of childbearing potential, have a negative pregnancy test on the day of surgery per standard of care
* Be at least 18, but not more than 80 years of age
* Have an ASA risk class of I, II, or III according to the American Society of Anesthesiologists (ASA).
* Have the ability to read and understand the study procedures and the use of the pain scales. Must have the ability to communicate meaningfully with the Study Investigator and staff.
* Be free of other physical, mental, or medical conditions, which in the opinion of the Investigator, makes study participation inadvisable.

Exclusion Criteria:

* Subjects requiring daily opioids equivalent to greater than 40 mg oxycodone for over 2 weeks prior to the study.
* Has significant preexisting pulmonary (respiratory/breathing) disease, diaphragmatic paralysis or history of phrenic nerve injury (problems with the diaphragm causing breathing difficulties).
* Has significant medical disease(s), laboratory abnormalities or condition(s) that in the Investigator's judgment could compromise the subject's welfare, ability to communicate with the study staff, complete study activities, or would otherwise contraindicate study participation.
* Has known significant hypersensitivity to opioids, Ropivacaine, or the inactive ingredients (excipients) of the study medications.
* Has known or suspected history of alcohol or drug abuse or dependence within the previous 2 years.
* Has clinically significant liver disease, or other condition (e.g., alcoholism, cirrhosis, or hepatitis) based on medical history and examination.
* Has participated in another clinical Study (investigational or marketed product within 30 days of surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hartrick, MD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospitals, Troy, Michigan

REFERENCES:
- [Result] Hartrick CT, Tang YS, Siwek D, Murray R, Hunstad D, Smith G. The effect of initial local anesthetic dose with continuous interscalene analgesia on postoperative pain and diaphragmatic function in patients undergoing arthroscopic shoulder surgery: a double-blind, randomized controlled trial. BMC Anesthesiol. 2012 Mar 23;12:6. doi: 10.1186/1471-2253-12-6. PMID 22443231

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were identified from the surgical schedule. Subjects consented using the most current IRB-approved consent form. Informed consent were administered in the pre-operative suites prior to receiving any treatment.
  Recruitment started after approval was obtained from the IRB. Recruitment period was Jan 2009 to Dec 2009.
Pre-assignment Details: Subjects were screened per protocol, those that met all inclusion criteria and did not meet any exclusion criteria were randomized per protocol.
Groups:
- Ropivacaine 5 mL: Initial Bolus 0f 5 ml Ropivacaine 0.75% administered as interscalene peripheral nerve block prior to surgical procedure performed with ultrasound guidance followed by a continuous infusion of Ropivacaine 0.2% using the Stryker Pain Pump II with the following setting: 3 ml bolus/demand, 4ml/hr continuous infusion with a 20 min lock-out.
- Ropivacaine 10 mL: Initial Bolus 0f 10 ml Ropivacaine 0.75% administered as interscalene peripheral nerve block prior to surgical procedure performed with ultrasound guidance followed by a continuous infusion of Ropivacaine 0.2% using the Stryker Pain Pump II with the following setting: 3 ml bolus/demand, 4ml/hr continuous infusion with a 20 min lock-out.
- Ropivacaine 20 mL: Initial Bolus 0f 20 ml Ropivacaine 0.75% administered as interscalene peripheral nerve block prior to surgical procedure performed with ultrasound guidance followed by a continuous infusion of Ropivacaine 0.2% using the Stryker Pain Pump II with the following setting: 3 ml bolus/demand, 4ml/hr continuous infusion with a 20 min lock-out.
Period: Overall Study
Arm/Group | Ropivacaine 5 mL | Ropivacaine 10 mL | Ropivacaine 20 mL
Started | 12 | 12 | 12
PACU (Within 8 Hours) | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine 5 mL | Ropivacaine 10 mL | Ropivacaine 20 mL | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 36
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 11
  Male | 7 | 9 | 9 | 25
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Pain Measurements Via Numeric Pain Rating Scales (NRS)
Description: Pain was reported via NRS ranging from 0 (no pain) to 10 (worst pain imaginable)
Time Frame: Discharge, 24 h, 48h, 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ropivacaine 5 mL | Ropivacaine 10 mL | Ropivacaine 20 mL
Number analyzed (Participants) | 12 | 12 | 12
units on a scale
  NRS at Discharge | 2.67 [0.61 to 4.71] | 1.58 [-0.18 to 3.35] | 0.62 [-0.26 to 1.49]
  NRS at 24 hours post discharge | 3.67 [2.03 to 5.30] | 3.33 [1.57 to 5.10] | 2.54 [1.09 to 3.99]
  NRS at 48 hours post discharge | 2.67 [1.08 to 4.25] | 2.08 [0.66 to 3.50] | 2.15 [0.92 to 3.38]
  NRS at 12 weeks post discharge (n=11, 12, 12) | 1.5 [0.50 to 2.50] | 2.42 [0.55 to 4.28] | 1.15 [0.42 to 1.89]

2. Primary Outcome: Change in Diaphragmatic Displacement From Baseline to Post-surgery
Description: Diaphragm displacement from exhale to inhale. The baseline diaphragm measurement was obtained pre-operatively before the block was administered prior to surgery. This was again measured post-operatively before the patient's discharge from the Post-anesthesia Care Unit.
Time Frame: Baseline, Post anesthesia care unit (PACU) - within 8 hours
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Ropivacaine 5 mL | Ropivacaine 10 mL | Ropivacaine 20 mL
Number analyzed (Participants) | 12 | 12 | 12
percent change
  % change in diaphragm displacement ipsilateral | 66 [43 to 88] | 60 [21 to 98] | 65 [45 to 86]
  % change in diaphragm displacement contralateral | -28 [-45 to -10] | -56 [-139 to 26] | -39 [-114 to 36]

3. Secondary Outcome: Percentage of Participants Who Considered the Analgesic Technique "Helpful" or "Extremely Helpful"
Description: Participants were asked to rate the helpfulness of their infusion:
  1. extremely harmful
  2. harmful
  3. neutral
  4. not harmful, but not helpful
  5. helpful
  6. extremely helpful
Time Frame: at 24 and 48 hours after discharge from the hospital
Measure: Number; unit: percentage of participants
Arm/Group | Ropivacaine 5 mL | Ropivacaine 10 mL | Ropivacaine 20 mL
Number analyzed (Participants) | 12 | 12 | 12
percentage of participants
  Percentage of participants at 24 hours | 83 | 83 | 92
  Percentage of participants at 48 hours | 83 | 75 | 85

4. Secondary Outcome: Functional Outcome - Simple Shoulder Test (SST)
Description: At baseline and again at 12 weeks subjects completed the Simple Shoulder Test. This test is a series of 12 (yes/no) questions. Participants get 1 point if they answer yes (they can perform the task) and 0 if they answer no. Total possible range is from 0-12. This has been shown to be a valid, reliable and consistent for subjects up to and including 60 years of age when similar injuries (rotator cuff dysfunction) are assessed.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- All Study Participants: All study participants who received Interscalene block (ISB) using 5-20 mL of local anesthetic.
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
units on a scale
  SST at Baseline (n=36) | 6.3 [5.1 to 7.5]
  SST at 12 weeks (n=35) | 8.2 [7.3 to 9.2]

ADVERSE EVENTS:
Arm/Group | Ropivacaine 5 mL | Ropivacaine 10 mL | Ropivacaine 20 mL
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes